CLINICAL TRIAL: NCT02865525
Title: QUILAM : Development and Validation of a Self-administered QUestionnaire to Identify Levers of Adhesion Behavior to Patient's Medication in Order to Adapt the Educational Monitoring
Brief Title: Development and Validation of a Self-administered QUestionnaire to Identify Levers of Adhesion Behavior to Patient's Medication in Order to Adapt the Educational Monitoring.
Acronym: QUILAM
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC14.084
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Patient Education as Topic; Surveys and Questionnaires; Medication Adherence; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus, Type 2; Heart Failure
Keywords: Surveys and Questionnaires; Patient Education as Topic; Medication Adherence; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus, Type 2; Heart failure
MeSH Terms: conditions — Medication Adherence; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus, Type 2; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Medication non-adherence is an economic problem and a major public health challenge. Factors influencing medication adherence can be modelled according to five dimensions: disease, medication, patient and its close relatives, demographic and socioeconomic factors and health care system. A tool is needed to qualify medication adherence in order to adapt tailored support for individual patients to promote and optimize adherence to therapy.

The objective of this work is to present the preliminary results of QUILAM project which is divided into 3 phases: 1. Development of a tool to assess barriers to medication adherence in chronic patient (COPD, Heart failure, Type 2 diabetes) ; 2. Validation of the instrument (especially against clinical criteria) ; 3. Evaluation of the sensitivity of the tool during educational interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patient with at least one of the following pathologies: diabetes type II, COPD, heart failure
* person available for a follow-up of 1 year
* Affiliated to the social security or recipient of such a regime

Exclusion Criteria:

* Persons referred to in articles L1121-5 and L1121-8 in the french public health code
* Patient who do not speak french

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: targeted pathologies: type 2 diabetes heart failure Chronic obstructive pulmonary disease
Sampling Method: Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Number of events 'hospitalization and death' for 2 patient groups defined through the questionnaire QUILAM score | 12 month

SECONDARY OUTCOMES:
Feasibility and acceptability of the questionnaire (duration / missing data) | 12 month
Reliability over time of the questionnaire (test-retest J0 - J15) | 12 month
External construct validity (Girerd, SatMedQ, BMQ) | 12 month
Number of clinical events for 2 patient groups | 12 month
Number of events 'hospitalization and death' for 2 patient groups separate with different cut off | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Benoît ALLENET, PharmD, PHD, Study Director — TIMC-IMAG UMR 5525 / ThEMAS, University Grenoble-Alpes/ Grenoble University Hospital, Grenoble, France/; Aurelie Gauchet, PHD, Study Director — Inter-University Laboratory of Psychology (LIP), University Grenoble-Alpes, Grenoble, France
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No